CLINICAL TRIAL: NCT00471445
Title: Assessment of Topical Treatment Response With Amitriptyline and Ketamine: Combination Trial in Chemotherapy Peripheral Neuropathy (ATTRACT-CPN)
Brief Title: Topical Amitriptyline and Ketamine Cream in Treating Peripheral Neuropathy Caused by Chemotherapy in Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gary Morrow (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Gary Morrow, Director, URCC NCORP Research Base, University of Rochester NCORP Research Base
Organization: University of Rochester (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CDR0000543103; U10CA037420 (NIH); URCC-0605 (Other: NCI/DCP); URCC07004 (Other: University of Rochester)
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Results first posted 2015-06-10 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-10

CONDITIONS: Neurotoxicity; Pain; Peripheral Neuropathy; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; pain; neurotoxicity; peripheral neuropathy
MeSH Terms: conditions — Neurotoxicity Syndromes; Pain; Peripheral Nervous System Diseases | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ketamine/amitriptyline NP-H cream (Experimental): Patients apply 4 grams amitriptyline (4%) and ketamine (2%) hydrochloride topical analgesic cream twice daily to areas of pain, numbness, or tingling in the hands and/or feet.
  Interventions: Drug: ketamine/amitriptyline NP-H cream
- Placebo Cream (Placebo Comparator): Patients apply a placebo cream twice daily to areas of pain, numbness, or tingling in the hands and/or feet.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: ketamine/amitriptyline NP-H cream — Subjects were instructed to apply up to, but not exceeding, 4 g of ketamine/amitriptyline NP-H cream two times per day to each area with pain, numbness, and/or tingling. A measuring device was provided to assist in dispensing the proper amount of the cream.
  Other Names: EpiCept NP-1
  Arms: ketamine/amitriptyline NP-H cream
Other: placebo — Applied topically
  Arms: Placebo Cream

SUMMARY:
RATIONALE: Topical cream containing amitriptyline and ketamine may help relieve pain, numbness, tingling, and other symptoms of peripheral neuropathy. It is not yet known whether topical amitriptyline and ketamine cream is more effective than a placebo in treating peripheral neuropathy caused by chemotherapy.

PURPOSE: This randomized phase III trial is studying the side effects and how well topical amitriptyline and ketamine cream work compared with a placebo in treating peripheral neuropathy caused by chemotherapy in patients with cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the analgesic properties and safety of topical amitriptyline and ketamine hydrochloride cream vs placebo in cancer patients with chemotherapy peripheral neuropathy (CPN) who have received taxanes or other cancer chemotherapy agents.

OUTLINE: This is a multicenter, double-blind, randomized, placebo-controlled study. Patients are stratified according to Community Clinical Oncology Program (CCOP) site. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients apply amitriptyline and ketamine hydrochloride topical analgesic cream twice daily to areas of pain, numbness, or tingling in the hands and/or feet.
* Arm II: Patients apply a placebo cream twice daily to areas of pain, numbness, or tingling in the hands and/or feet.

In both arms, treatment continues for 6 weeks in the absence of disease progression or unacceptable toxicity. Patients may continue treatment for up to a total of 12 weeks.

Patients complete a peripheral neuropathy intensity and quality of sleep diary daily. Patients also complete the European Organization for Research and Treatment of Cancer Quality of Life-Chemotherapy-Induced Peripheral Neuropathy (EORTC-CIPN20) to assess change in sensory score and the Brief Pain Inventory and Hospital Anxiety and Depression Scale to assess health-related quality of life in week 3 and 6. The Vulnerable Elders Survey (VES-13) is administered at baseline to assess level of physical activity and the University of Rochester Cancer Center (URCC) symptom inventory is administered to track other potentially important symptoms. The Patient Global Impression of Change Questionnaire is administered in week 6 to assess the patient's overall assessment of change since beginning treatment, including changes in pain, side effects, functional status, and overall satisfaction with treatment.

PROJECTED ACCRUAL: A total of 462 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* History of cancer
* Pain, numbness, or tingling in the hands or feet beginning in association with a cancer chemotherapy agent (taxane or other chemotherapeutic agent) and persisting for at least 28 days following the conclusion of chemotherapy

  * Pain, numbness, or tingling can be assessed 28 days or more after the conclusion of chemotherapy
  * An average score of ≥ 4 for the 7 daily ratings of the baseline week on the 11-point rating scale of peripheral neuropathy associated with chemotherapy, with a minimum of 5 daily diary ratings completed during the baseline week
* No preexisting or history of peripheral neuropathy due to any cause other than chemotherapy (e.g., hereditary, alcohol, or diabetes)
* Patients with stable systemic metastases and/or bone involvement AND has not received chemotherapy within 3 months of screening assessment are eligible

  * Patients receiving ongoing treatment with non-chemotherapy agents (e.g., monoclonal antibodies or hormonal treatment) allowed
* No concurrent active chemotherapy in the adjuvant setting or for progressive systemic disease

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Creatinine ≤ 2 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to adequately understand English
* No allergy or hypersensitivity to ketamine hydrochloride or amitriptyline or any of the components of study drug
* No clinically significant illness (e.g., endocrine, cardiac, hepatic, renal, neurologic, hematologic, or skeletal illness) that, in the investigator's clinical judgment, could interfere with the efficacy or safety assessments in this study
* No glaucoma or recurrent urinary retention
* No clinically significant depression or dementia that, in the opinion of the investigator, may interfere with a patient's adherence to the study protocol and/or the accurate and consistent reporting of CPN
* No open skin lesions in the area where the cream is to be applied
* No HIV positivity

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 30 days since prior unapproved experimental drugs or biological agents
* No prior topical treatment, nerve blocks, implantable therapy, peripheral nerve or spinal cord stimulation, or neurosurgical procedure for chemotherapy-related peripheral neuropathy (CPN)
* No prior exposure to a peripheral neurotoxin other than chemotherapy
* No concurrent medications (e.g., phenytoin) known to be associated with sensory neuropathy
* No concurrent selective serotonin reuptake inhibitors (e.g., fluoxetine, paroxetine, or sertraline), which inhibit CP450 2D6, unless the patient is being treated for depression or another psychiatric disorder and, in the investigator's judgment, the patient's participation in the study can be permitted given the minimal systemic levels of amitriptyline found within the cream
* No concurrent monoamine oxidase inhibitors, barbiturates, anticholinergic agents, or sympathomimetic drugs, including epinephrine combined with local anesthetics

  * Oral inhalers that include any of the drugs listed above are allowed
* Concurrent opioid analgesics, tricyclic or dual reuptake inhibitor antidepressants, or gabapentin or pregabalin for CPN, or benzodiazepines for sleep allowed, provided dose has been stable for ≥ 2 weeks and the following are true:

  * Gabapentin dose ≤ 1,800 mg per day
  * Pregabalin dose ≤ 300 mg per day
  * Opioid analgesic dose ≤ 60 mg oxycodone hydrochloride equivalent per day
  * Tricyclic antidepressant dose ≤ 75 mg amitriptyline equivalent per day
  * Duloxetine dose ≤ 60 mg per day
  * Venlafaxine dose ≤ 150 mg per day
  * Tramadol dose ≤ 200 mg per day
* Concurrent adjunctive analgesic therapy, such as acupuncture, biofeedback, or herbal preparations, allowed provided dose has been stable for ≥ 2 weeks

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2007-10; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Supriya Mohile, MD, Study Chair — James P. Wilmot Cancer Center
Locations (17):
- United States (17):
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin

REFERENCES:
- [Derived] Gewandter JS, Mohile SG, Heckler CE, Ryan JL, Kirshner JJ, Flynn PJ, Hopkins JO, Morrow GR. A phase III randomized, placebo-controlled study of topical amitriptyline and ketamine for chemotherapy-induced peripheral neuropathy (CIPN): a University of Rochester CCOP study of 462 cancer survivors. Support Care Cancer. 2014 Jul;22(7):1807-14. doi: 10.1007/s00520-014-2158-7. Epub 2014 Feb 16. PMID 24531792

RESULTS

PARTICIPANT FLOW:
Groups:
- Amitriptyline and Ketamine Hydrochloride Topical Analgesic cr: Patients apply amitriptyline and ketamine hydrochloride topical analgesic cream twice daily to areas of pain, numbness, or tingling in the hands and/or feet.
  ketamine/amitriptyline NP-H cream: Applied topically
Period: Overall Study
Arm/Group | Amitriptyline and Ketamine Hydrochloride Topical Analgesic cr | Placebo Cream
Started | 229 | 233
Completed | 227 | 231
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Ineligible | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: The number of 458 does not include 2 subjects from the Placebo cream and 2 subjects from the Amitriptyline and ketamine hydrochloride topical analgesic cream group who did not provide baseline data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Amitriptyline and Ketamine Hydrochloride Topical Analgesic cr | Placebo Cream | Total
Number analyzed (Participants) | 227 | 231 | 458
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (10.5) | 60.6 (10.0) | 60.7 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 156 | 171 | 327
  Male | 71 | 60 | 131
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 220 | 224 | 444
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 18 | 38
  White | 199 | 206 | 405
  More than one race | 8 | 7 | 15
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 227 | 231 | 458
Education [Number; unit: participants]
  Completed graduate training | 28 | 19 | 47
  Standard college or university (4 years) | 53 | 55 | 108
  Partial college training (<4 years) | 76 | 80 | 156
  High school graduate | 63 | 65 | 128
  Not high school educated | 7 | 12 | 19
Marital status [Number; unit: participants]
  Married | 165 | 160 | 325
  Divorced | 20 | 25 | 45
  Separated | 2 | 3 | 5
  Single | 23 | 21 | 44
  Widowed | 17 | 22 | 39
Previous treatment [Number; unit: participants] — Sum of participants in each treatment category will not sum to the overall number of baseline participants since participants may belong in multiple categories.
  participants
    Previous surgery | 198 | 195 | 393
    Previous chemotherapy | 227 | 231 | 458
    Previous radiation therapy | 114 | 109 | 223
Site [Number; unit: participants] — Sum of participants in each site category will not sum to the overall number of baseline participants since participants may belong in multiple categories.
  participants
    Hematologic | 24 | 18 | 42
    Head and neck | 7 | 5 | 12
    Lung | 12 | 23 | 35
    GI | 55 | 69 | 124
    Genitourinary tract | 15 | 9 | 24
    Gynecologic | 15 | 16 | 31
    Breast | 96 | 88 | 184
    Skin | 1 | 1 | 2
    Melanoma | 0 | 1 | 1
    Soft tissue sarcoma | 2 | 1 | 3
    Bone and cartilaginous | 2 | 0 | 2
    Cardiac | 0 | 1 | 1
    Other | 5 | 4 | 9
Regimen [Number; unit: participants]
  Taxanes | 126 | 120 | 246
  Non-Taxane | 101 | 111 | 212

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Daily Peripheral Neuropathy Intensity Score From Baseline to Week 6 in Patients Treated With Amitriptyline and Ketamine Hydrochloride vs Placebo
Description: Cancer survivors who completed chemotherapy at least 1 month prior and had Chemotherapy Induced Peripheral Neuropathy (CIPN) (greater than or equal to 4 out of 10) were enrolled. CIPN was assessed using average scores from a 7-day daily diary that asks patients to rate the average "pain, numbness, or tingling in their hands and feet over the past 24 hours" on an 11-point numeric rating scale at baseline and 6 weeks post intervention. CIPN ranges from 0 (no pain) to 10 (worst possible pain).
Time Frame: Week 6 - Baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Ketamine/Amitriptyline NP-H Cream: Patients apply amitriptyline and ketamine hydrochloride topical analgesic cream twice daily to areas of pain, numbness, or tingling in the hands and/or feet.
  ketamine/amitriptyline NP-H cream: Applied topically
Arm/Group | Ketamine/Amitriptyline NP-H Cream | Placebo Cream
Number analyzed (Participants) | 227 | 231
units on a scale
  Baseline | 6.55 [6.35 to 6.76] | 6.47 [6.28 to 6.66]
  Week 6 | 4.93 [4.59 to 5.27] | 5.19 [4.89 to 5.49]
Statistical Analysis 1: Comparison: Ketamine/Amitriptyline NP-H Cream vs Placebo Cream; Tested at the two-sided 0.05 significance level; Test type: Superiority or Other; p = 0.363, ANCOVA; Mean Difference (Final Values) = -0.174, 95% CI 2-sided [-0.548 to 0.201], Standard Error of Mean 0.190

ADVERSE EVENTS:
Arm/Group | Amitriptyline and Ketamine Hydrochloride Topical Analgesic cr | Placebo Cream
Serious Adverse Events (participants affected / at risk) | 4/227 | 4/231
Other Adverse Events (participants affected / at risk) | 147/227 | 158/231
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amitriptyline and Ketamine Hydrochloride Topical Analgesic cr (N=227) | Placebo Cream (N=231)
Allergic Rhinitis (Immune system disorders) | 0 | 1
Arrythmia recurrence - pacemaker placed (Cardiac disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Sensory Neuropathy (Nervous system disorders) | 1 | 0
Pain in ribs (Musculoskeletal and connective tissue disorders) | 1 | 0
Skin Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Open Heart Surgery (Cardiac disorders) | 1 | 0
Vaginal Bleeding (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amitriptyline and Ketamine Hydrochloride Topical Analgesic cr (N=227) | Placebo Cream (N=231)
Anorexia (Metabolism and nutrition disorders) | 3 | 1
Chills (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Dizziness (Ear and labyrinth disorders) | 2 | 3
Drymouth (Metabolism and nutrition disorders) | 1 | 0
Fatigue (General disorders) | 8 | 11
Fever (Infections and infestations) | 3 | 4
Tinnitus (Ear and labyrinth disorders) | 2 | 1
Hotflashes (General disorders) | 1 | 0
Insomnia (General disorders) | 5 | 7
Liver enzymes (Hepatobiliary disorders) | 2 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Infection - Herpes Zoster (Infections and infestations) | 2 | 1
Edema - Upper Extremities (Skin and subcutaneous tissue disorders) | 2 | 1
Edema - Lower Extremities (Skin and subcutaneous tissue disorders) | 1 | 4
Burning Sensation (Skin and subcutaneous tissue disorders) | 4 | 3
Rash - NOS (Skin and subcutaneous tissue disorders) | 2 | 7
Rash - Lower Extremities (Skin and subcutaneous tissue disorders) | 5 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 4 | 1
Skin Ulcerations (Skin and subcutaneous tissue disorders) | 1 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 2 | 1
Feeling of Tightness / Flusing in Feet (Skin and subcutaneous tissue disorders) | 2 | 0
Allergic Rhinitis (Immune system disorders) | 5 | 2
Red and Crusty Eye (Immune system disorders) | 1 | 0
Nasal Congestion (Immune system disorders) | 1 | 3
Hypertension (Cardiac disorders) | 5 | 5
Cardiac Arrythmia (Cardiac disorders) | 1 | 1
Increased Heart Rate (Cardiac disorders) | 2 | 1
Congestive Heart Failure (Cardiac disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbumin (Metabolism and nutrition disorders) | 1 | 1
Hypotension (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesium (Metabolism and nutrition disorders) | 0 | 1
Diabetes (Endocrine disorders) | 0 | 2
Hypothyroidism (Endocrine disorders) | 2 | 1
Hyperglycemia (Endocrine disorders) | 6 | 2
Hypercholestremia (Endocrine disorders) | 0 | 1
Hyperlipidemia (Endocrine disorders) | 1 | 0
Urinary Tract Infection (Reproductive system and breast disorders) | 2 | 3
Benign Prostate Hyperplasia (Reproductive system and breast disorders) | 0 | 1
Bladder Spasms, Occasional (Reproductive system and breast disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 3 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Head Cold (Infections and infestations) | 1 | 2
Otitis Media (Infections and infestations) | 1 | 0
Headache (General disorders) | 4 | 3
Anxiety (Psychiatric disorders) | 1 | 6
Depression (Psychiatric disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 2 | 7
Vomiting (Gastrointestinal disorders) | 2 | 4
Abdominal Pain (Gastrointestinal disorders) | 3 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 6
Dysphagia (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 4
Constipation (Gastrointestinal disorders) | 1 | 4
GI Fistula (Gastrointestinal disorders) | 1 | 0
GERD (Gastrointestinal disorders) | 2 | 0
Mucositis (Gastrointestinal disorders) | 1 | 1
Black Tarry Stool (Gastrointestinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Migraine (Nervous system disorders) | 3 | 1
Neuropathy (Nervous system disorders) | 6 | 8
Ataxia (Nervous system disorders) | 1 | 0
Cramps (Nervous system disorders) | 2 | 2
Restless Leg Syndrome (Nervous system disorders) | 4 | 0
Pain Lower Extremities (Musculoskeletal and connective tissue disorders) | 5 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 11
Pain in Joint (Musculoskeletal and connective tissue disorders) | 5 | 4
Pain Upper Extremities (Musculoskeletal and connective tissue disorders) | 2 | 4
Pain in Bone (Musculoskeletal and connective tissue disorders) | 3 | 0
Pain in Knee (Musculoskeletal and connective tissue disorders) | 4 | 2
Pain in Head / Neck (Musculoskeletal and connective tissue disorders) | 4 | 3
Pain in Back (Musculoskeletal and connective tissue disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
Since ketamine and amitriptyline are both analgesics, it is possible that the effects of the ketamine plus amitriptyline-containing creams may have been diluted when all three neuropathy symptoms were assessed together.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No